CLINICAL TRIAL: NCT07111702
Title: Prophylactic Antibiotics in Groin Hernioplasty: A Prospective Cohort Study on the Prevention of Surgical Site Infection
Brief Title: Prophylactic Antibiotics in Groin Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Collaborators: Al-Gumhori Teaching Hospital (Unknown)
Responsible Party: Principal Investigator, Haitham Mohammed Jowah, Lecturer, Sana'a University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-Hernia-001
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Surgical Site Infection; Groin Hernia; Hernioplasty
Keywords: Antibiotic Prophylaxis; Wound Infection; Risk Factors
MeSH Terms: conditions — Surgical Wound Infection; Hernia, Inguinal; Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic Group (Experimental): Patients received a single intravenous dose of cefazolin (2 g) 30-60 min prior to skin incision.
  Interventions: Drug: Cefazolin
- No Antibiotic Group (No Intervention): Patients did not receive antibiotic prophylaxis.

INTERVENTIONS:
Drug: Cefazolin — A single 2g intravenous dose administered once before surgery.
  Arms: Antibiotic Group

SUMMARY:
The role of prophylactic antibiotics in preventing surgical site infections (SSI) for clean procedures like groin hernia repair remains controversial. This study aimed to evaluate the association between antibiotic prophylaxis and SSI rates in a real-world clinical setting and to identify independent risk factors for SSI. The study prospectively followed 100 male patients undergoing elective open groin hernioplasty. Patients were categorized based on the surgeon's decision into two groups: those who received a single dose of intravenous cefazolin (Antibiotic Group) and those who did not (No Antibiotic Group). The main outcome was the rate of SSI within 30 days of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 17-80 years) undergoing primary open groin hernioplasty.
* Provided written informed consent.

Exclusion Criteria:

* Recurrent, emergency, or complicated (e.g., incarcerated, strangulated) hernias.
* Laparoscopic repairs.
* Known immunosuppression, ongoing antibiotic therapy, or a known allergy to cefazolin.
* Refusal to participate.

Ages: 17 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection (SSI) | Within 30 days post-surgery
  The rate of surgical site infection diagnosed within 30 days of surgery, based on Centers for Disease Control and Prevention (CDC) clinical criteria (e.g., purulent discharge, erythema, localized pain or swelling).

SECONDARY OUTCOMES:
Independent Risk Factors for Surgical Site Infection (SSI) | From baseline through 30 days post-surgery
  Identification of baseline and operative variables independently associated with the development of SSI. This was assessed using a multivariable logistic regression model to calculate adjusted odds ratios for factors such as high Body Mass Index (BMI), prolonged operative time, and high American Society of Anesthesiologists (ASA) score.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Mohammed Gilan, Asssociate Professor, Principal Investigator — Faculty of Medicine and Health Sciences, Sana'a University
Locations (1):
- Al-Gumhori Teaching Hospital, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article will be made available after publication. This includes data on baseline characteristics, group allocation, and the primary outcome.
Time Frame: Data will be available beginning 3 months after article publication and the access period will remain open for 5 years.
Access Criteria: Data will be made available to qualified researchers for meta-analysis or other secondary analyses. Researchers must submit a methodologically sound proposal to the corresponding author at h.jowah@su.edu.ye. A signed data access agreement will be required.